CLINICAL TRIAL: NCT05357170
Title: Microbiome Dysfunction in Surgical Intensive Care Unit Survivors Subtitle: The Role of Brain-Bone Marrow-Gut Interaction Following Major Trauma Pathological Myeloid Activation After Sepsis and Trauma
Brief Title: Microbiome Dysfunction in Surgical Intensive Care Unit Survivors
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB202102863; R35GM140806 (NIH)
Record Dates: First submitted 2022-04-12; First posted 2022-05-02 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Sepsis, Trauma Injury
Keywords: Sepsis; Trauma; Microbiome
MeSH Terms: conditions — Sepsis; Accidental Injuries; Wounds and Injuries | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human oral sample, feces, and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Sepsis Survivors: Oral swab, saliva, and feces collected between 7 to 28 days of hospital admission and at 3 and 6 months post hospitalization. Telephone call at 12 months.
  Blood will be collected at time of first feces collection
  Interventions: Other: Human feces collection
- Healthy Control Population: One time collection of oral swab and saliva, feces, and blood upon enrollment used for comparison to identify microbial genes associated with persistent systemic inflammation in sepsis survivors.
  Interventions: Other: Human feces collection
- Trauma Survivor: Oral swab, saliva, and feces collected between 7 to 28 days of hospital admission and at 3 and 6 months post hospitalization. Telephone call at 12 months.
  Blood will be collected at time of first feces collection
  Interventions: Other: Human feces collection
- Traumatic Brain Injury (TBI): Oral swab, saliva, and feces collected at admission (day 1(+5)) and between 7 to 28 days of hospital admission and at 3 and 6 months post hospitalization. Telephone call at 12 months.
  Blood will be collected at time of first and second feces collection.
  Interventions: Other: Human feces collection
- Cardiopulmonary Bypass: Oral swab, saliva, and feces collected between 7 to 28 days of hospital admission and at 3 and 6 months post hospitalization. Telephone call at 12 months.
  Blood will be collected at time of first feces collection
  Interventions: Other: Human feces collection
- Major Vascular Surgery: Oral swab, saliva, and feces collected between 7 to 28 days of hospital admission and at 3 and 6 months post hospitalization. Telephone call at 12 months.
  Blood will be collected at time of first feces collection
  Interventions: Other: Human feces collection

INTERVENTIONS:
Other: Human feces collection — Oral swab and saliva, human feces collection and blood sampling
  Other Names: Blood sampling; Oral swab and saliva

SUMMARY:
Oral and gastrointestinal microbiome dysfunction has been demonstrated to be a culprit of various systemic dysfunctions in peripheries such as cardiovascular, nervous, endocrine and musculoskeletal systems. The topic of microbiome dysfunction after surgical intensive care admission is understudied but may be responsible for persistent systemic inflammation clinically observed in surgical intensive care patients. Therefore, the objective of this project is to investigate the oral and gut microbiome after the acute phase of sepsis, severe trauma injury, cardiopulmonary bypass, and major vascular surgery to compare with 108 age-matched healthy population controls

DETAILED DESCRIPTION:
The investigators hypothesize that alterations of the oral and gut microbiota will correlate with persistent systemic inflammation in surgical intensive care unit survivors compared to existing healthy population controls. This research group will collect oral and stool samples from 108 sepsis survivors, 108 trauma survivors, 108 cardiopulmonary bypass survivors, and major vascular surgery survivors (groups of ages 18-45, 46-64, and >65; male and female; n=18 per age + sex cohort) admitted to the surgical intensive care unit between day 7 and 28 of hospital admission, as well as 3 and 6 months after their intensive care unit hospitalization. The investigators will perform 16S rRNA DNA sequencing on the isolated bacterial DNA from these samples and bioinformatic analysis to determine microbiota alterations between time points and between surgical ICU survivor cohorts and a control cohort. In addition, the investigators will draw 20ml of blood to isolate plasma.

Trauma Subgroup for traumatic brain injury (TBI) pilot study: Our team will enroll 15 additional trauma injury patients with traumatic brain injury. This subgroup will have an added stool (if available) and blood sample collection after initial injury (+ 5 days). The additional sample will be compared to the sample collected at 14-21 days and follow up samples at 3 and 6 months. The results will be associated with Glasgow Outcome Scale Extended at 3 and 12 month time points and the recorded discharge Rancho Los Amigos scale score from the medical record. The specific aims will be: Aim 1 - define the impact of persistent systemic inflammation on the gastrointestinal microbiota in sepsis and trauma survivors and Aim 2 - identify microbial genes associated with persistent systemic inflammation in sepsis and trauma survivors compared to normal controls. Trauma Subgroup Aim: Pilot study to test the hypothesis that changes in the microbiome towards pathogenic microbe is associated with worsened outcomes in trauma injury patients with TBI (traumatic brain injury).

ELIGIBILITY:
Sepsis Population

Inclusion Criteria

1. Admission to the 46, 77, 87, 4 East, 4 West, or 24-5 ICUs where clinical care can be managed by the critical care organization guided by standard operating procedures.
2. Age ≥18 years
3. Meets Sepsis 3 criteria at time of sepsis diagnosis
4. Has remained in ICU for 14 days (+/- 7 days) following sepsis diagnosis.
5. Ability to obtain patient/LAR informed consent.
6. Is receiving adequate nutritional intake: oral or enteral nutrition.

Exclusion Criteria

1. Severe traumatic brain injury with unencumbered assessment of GCS equaling 3 on admission to intensive care unit
2. Refractory shock (i.e., patients who are expected to die within 12 hours).
3. Uncontrollable source of sepsis (e.g. irreversible disease state such as unresectable dead bowel).
4. Patient or patient's family are not committed to aggressive management of the patient's condition.
5. Known HIV infection with CD4 count <200 cells/mm3.
6. Organ transplant recipient on immunosuppressive agents.
7. Known pregnancy.
8. Prisoners.
9. Institutionalized patients j Inability to obtain informed consent.

k) Burn injury greater than 20% TBSA (total body surface area)

Trauma Population

Inclusion Criteria

1. All adults (age ≥18 to 54) require both:

a. Blunt and/or penetrating trauma patient with i. Hemorrhagic shock defined by:

1. Systolic BP (SBP) ≤ 90 mmHg or 2. Mean arterial pressure ≤ 65 mmHg or 3. Base deficit (BD) ≥5 meq or 4. Lactate ≥ 2 or 5. Active red blood cell or whole blood transfusion within 6 hours of arrival

b. Injury Severity Score (ISS) greater than or equal to 15

2. All adults (age 55 and older) require:

a. Either hemorrhagic shock defined by: i. Systolic BP (SBP) ≤ 90 mmHg or ii. Mean arterial pressure ≤ 65 mmHg or iii. Base deficit (BD) ≥5 meq or iv. Lactate ≥ 2 or v. Active red blood cell or whole blood transfusion within 6 hours of arrival

OR

b. Injury Severity Score (ISS) greater than or equal to 15. 3. Ability to obtain Informed Consent

Exclusion Criteria

1. Patients not expected to survive greater than 48 hours.
2. Prisoners.
3. Pregnancy.
4. Previous bone marrow transplantation.
5. Patients with End Stage Renal Disease.
6. Patients with any pre-existing hematological disease (e.g. hemochromatosis, myelodysplastic syndrome, hematologic cancers)
7. Burn injury greater than 20% TBSA
8. Severe traumatic brain injury with unencumbered assessment of GCS equaling 3 on admission to intensive care unit.

Trauma TBI subgroup (15 participants)

Inclusion criteria will be:

1. Any adult age 18 or older with any traumatic bleed (intracerebral hemorrhage, subarachnoid hemorrhage, intraparenchymal hemorrhage, subdural hematoma, cerebral epidural hematoma) and any GCS (Glasgow Coma Score).

Exclusion criteria is the same used for the trauma cohort.

Cardiac-Surgery operation:

Inclusion Criteria:

1. Adult (>18 years age) patients undergoing open cardiac surgery
2. Ability to obtain patient informed consent
3. was placed on cardiopulmonary bypass at their initial operation at UF Health

Exclusion Criteria:

1. Inability to obtain informed consent,
2. Pregnancy
3. Evidence of multi-organ failure on presentation
4. Patients with any pre-existing hematological disease (e.g. hemochromatosis, myelodysplastic syndrome, hematologic cancers
5. Prisoners
6. Previous bone marrow transplantation
7. Burn injury greater than 20% TBSA

Open abdominal vascular operation:

Inclusion Criteria:

1. Adult (>18 years age) patients undergoing open abdominal vascular surgery
2. Ability to obtain patient informed consent,

Exclusion Criteria:

1. Inability to obtain informed consent,
2. Pregnancy
3. Evidence of multi-organ failure on presentation
4. Patients with any pre-existing hematological disease (e.g. hemochromatosis, myelodysplastic syndrome, hematologic cancers
5. Prisoners
6. Previous bone marrow transplantation.
7. Burn injury greater than 20% TBSA

Healthy Control

Inclusion criteria will be:

1. All adults (age ≥18)
2. Ability to obtain Informed Consent prior to blood collection.

Exclusion Criteria will be:

1. Current, chronic steroid use
2. Pregnancy
3. Current or recent (within 7 days) use of antibiotics.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to surgical intensive care units who screen positive for sepsis, have severe trauma injury, undergo cardiopulmonary bypass or major vascular surger and are being treated by our standard-of care ICU protocols are candidates for the study. Healthy adult volunteers will provide reference control samples.
Sampling Method: Probability Sample
Enrollment: 468 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Determine the impact of persistent systemic inflammation on oral and gastrointestinal microbiota in surgical ICU survivors & identify microbial genes associated with persistent systemic inflammation of surgical ICU survivors compared to normal controls. | through study completion, an average of 6 months
  Identify oral and gut microbiome dysfunction through Microbial Taxonomic Analysis and Meta-transcriptomic Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Philip Efron, MD, Principal Investigator — UF COM Department of Surgery
Locations (1):
- UF Health at Shands Hospital, Gainesville, Florida, United States